CLINICAL TRIAL: NCT04798326
Title: A Single Center, Randomized, Double-blind , Single-dose, and Parallel Group Study to Compare the Pharmacokinetic, Safety and Pharmacodynamic of MW032 and Xgeva® in Healthy Adults
Brief Title: Comparing of the Pharmacokinetic, Pharmacodynamic, Safety and Immunogenicity of MW032 and Xgeva® in Healthy Adults
Acronym: MW032
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW032-2019-CP101
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Bone Tumor
Keywords: Denosumab; Biosimilar
MeSH Terms: conditions — Bone Neoplasms | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MW032 (Experimental): MW032 injection (120mg) by subcutaneous injection once on the first day of treatment.
  Interventions: Drug: MW032
- Xgeva® (Active Comparator): Xgeva® injection (120mg) by subcutaneous injection once on the first day of treatment.
  Interventions: Drug: Xgeva®

INTERVENTIONS:
Drug: MW032 — Subjects would receive a single 120mg (1.7 mL) of MW032 through subcutaneous injection, on the first day of treatment.
  Arms: MW032
Drug: Xgeva® — Subjects would receive a single 120mg (1.7 mL) of Xgeva® through subcutaneous injection, on the first day of treatment.
  Arms: Xgeva®

SUMMARY:
A randomized, double-blind and parallel group study to compare the pharmacokinetic, safety and pharmacodynamic of MW032 and Xgeva® in healthy adults.

DETAILED DESCRIPTION:
This is a phase I, single center, randomized, double-blind and parallel group clinical trial.

The primary objective is to assess the pharmacokinetic similarity of single and subcutaneous injections of MW032 and Xgeva® in healthy volunteers.

The secondary objective are to assess the Clinical safety and immunogenicity similarity of single and subcutaneous injections of MW032 and Xgeva® in healthy volunteers.

At the same time, preliminary evaluate the pharmacodynamic similarity between MW032 and Xgeva®.

Subjects would receive a single 120mg（1.7mL）of MW032 or Xgeva® through subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old (including 18 and 65 years old), healthy male subjects.
* Body mass index (BMI) within the range 19-28kg/m2.
* History, physical examination, laboratory tests and test related items of inspection were normal or mildly abnormal clinically insignificant.
* Volunteered to participate in this clinical trial, capable of giving written informed consentan.
* The subject (including the subject's partner) takes effective contraceptive measures.

Exclusion Criteria:

* Nervous/mental, respiratory system, cardiovascular system, digestive system, blood and lymphatic system, endocrine system, skeletal and muscular system diseases, liver and kidney dysfunction, or any other diseases and physiological conditions that may affect the results of the study.
* Occurred or suffering from osteomyelitis or ONJ (mandibular necrosis) previously.
* Clinical laboratory abnormalities of clinical significance, or other clinical findings suggest clinically significant following diseases (including, but not limited to the gastrointestinal tract, kidney, liver, nerve, blood, endocrine, cancer, lung, immune, mental or cardiovascular disease).
* Subject has viral hepatitis (including hepatitis B and hepatitis C), AIDS antibodies, and Treponema pallidum antibodies.
* Those who have used the following drugs within 1 month or 5 half-lives (whichever is longer) before participating in this study, including but not limited to: estrogen-containing contraceptives, bisphosphonates, fluoride, hormone replacement Treatment (ie tibolone, estrogen, estrogen-like compounds, such as raloxifene), calcitonin, strontium, parathyroid hormone or its derivatives, vitamin D supplements (>1000 IU/day), corticosteroids (inhaled or topical corticosteroids can be used 2 weeks before enrollment), anabolic hormone drugs, calcitriol, diuretics.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-t ) | Day0-Day161
Maximum serum concentration (Cmax) | Day0-Day161

SECONDARY OUTCOMES:
Adverse events(AE) | Day0-Day161
  The adverse medical events that occur after the clinical trial subjects receive the test drug do not necessarily have a causal relationship with the treatment.
serum CTX1 | Day0-Day161
  CTX1 is a serum type I collagen C-terminal peptide to detect the bone metastasis events.

CONTACTS AND LOCATIONS:
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China